CLINICAL TRIAL: NCT01980277
Title: A Prospective, Multicentre, Uncontrolled, Phase Ib/II Study of LY2780301 in Combination With Weekly Paclitaxel in HER2-negative Metastatic or Locally Advanced Breast Cancer in Patients With and Without PI3/AKT/S6 Pathway Activation. - TAKTIC-IPC 2012-008
Brief Title: Phase Ib/II Study of LY2780301 in Combination With Weekly PACLITAXEL in HER2-metastatic Breast Cancer
Acronym: TAKTIC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Drug development stopped
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAKTIC - IPC 2012-008
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LY2780301 + paclitaxel (Experimental): The following dose-levels will be investigated:
  * Continuous daily PO LY2780301 400 mg QD + weekly paclitaxel 70 mg/m²/week
  * Continuous daily PO LY2780301 400 mg QD + weekly paclitaxel 80 mg/m²/week
  * Continuous daily PO LY2780301 500 mg QD + weekly paclitaxel 80 mg/m²/week
  A dose reduction could be explored:
  - Continuous daily PO LY2780301 300 mg QD + weekly paclitaxel 70 mg/m²/week
  Interventions: Drug: LY2780301 + paclitaxel

INTERVENTIONS:
Drug: LY2780301 + paclitaxel — Continuous daily PO LY2780301 (400 mg, 500 mg or 300 mg) QD + weekly paclitaxel (70 or 80 mg/m²/week) for 21 days cycle until progression or toxicity

SUMMARY:
The overall rationale of this study evaluating tolerance and efficacy of LY2780301 in combination with paclitaxel in HER2-negative, inoperable locally advanced or metastatic breast cancer (MBC) is based on :

* the medical need in this population with either hormonal-resistant or unsensitive and/or rapidly progressive disease
* the preclinical evidences for involvement of PI3K/AKT pathway in tumor progression and drug resistance, including taxanes as well as its potential reversion by AKT inhibition
* the high level of frequency of PI3K/AKT activation in HER2-negative MBC
* the in vitro and in vivo preclinical activity of LY2780301, and its synergistic combination with various anticancer agents, including taxanes
* the favourable profile of tolerance of LY2780301 in phase I trial

Weekly paclitaxel is conventionally administered at 80 mg/m²/week and is a standard treatment in breast cancer (BC) As described above, LY2780301 500 mg once daily has been established as the RP2D in phase I single agent trial.

Evidence of pharmacodynamic activity was noted at 400-500 mg QD. Conservatively, the first dose level to be explored will be LY2780301 400 mg QD and paclitaxel 70 mg/m²/week.

DETAILED DESCRIPTION:
RATIONALE OF THE STUDY DESIGN

The purpose of this study will be:

1. to determine the recommended phase 2 dose (RP2D) for LY2780301 in combination with weekly paclitaxel in HER2-negative, inoperable locally advanced or MBC patients
2. to estimate the objective response rate (ORR) of the combination in first-line treated, HER2-negative, inoperable locally advanced or MBC patients. In addition, this study will assess the role of PI3K/AKT/S6 pathway activation as potential predictive factor for response to LY2780301 in this patient population.

This trial will be a phase Ib/II prospective, multicentre, open label, uncontrolled study.

Phase Ib will use a continuous reassessment method (CRM) design, allowing to reach safely and quickly the MTD and the RP2D of the combination, but ensuring the treatment of at least 18 patients to secure the tolerance profile.

Phase II will estimate antitumor activity in the overall patient population and in patients with activation of PI3K/AKT/S6 axis, allowing to examine its potential value as predictive biomarker

ELIGIBILITY:
Inclusion Criteria:

1. Female or male patients (≥ 18 years)
2. WHO/ECOG performance status ≤ 1 for phase Ib part, < 2 for phase II part
3. Patient with histologically confirmed inoperable locally advanced BC or MBC
4. Patient with tumor biopsy from metastatic tissue containing more than 50% tumor cells
5. Patient has known hormone receptor (ER/PR) status, positive and/or negative (local laboratory testing)
6. Patient has HER2-negative disease: IHC 0, 1 + or 2+ and/or in situ hybridization (FISH, CISH, SISH) negative (local laboratory testing)
7. Phase Ib: Patient has measurable or non-measurable disease according to RECIST 1.1 criteria only Phase II: Patient has measurable disease according to RECIST 1.1 criteria only
8. Patient has adequate bone marrow and organ function
9. Patient is able to swallow and retain oral medication
10. Negative serum pregnancy test within ≤ one week before first dose for childbearing potential women and for women < 12 months after the onset of menopause
11. Males and Females of childbearing potential (FCBP) must agree to use a reliable form of contraception or to practice complete abstinence from heterosexual intercourse during the study treatment (and 3 months after the end of treatment)
12. Life expectancy > 3 months
13. Affiliation to social security or beneficiary
14. Patient has signed the Informed Consent (ICF) prior to any screening procedures being performed

Exclusion criteria

1. Previous treatment with AKT or PI3K inhibitor
2. no previous cytotoxic treatment for metastatic or inoperable locally advanced disease (phase II part); Adjuvant/neoadjuvant therapy will be counted as prior line of therapy for metastatic/recurrent disease if the patient had a progression/recurrence within 6 months after completion of the therapy (12 months for taxane-based therapy). Previous hormonal treatment for metastatic or locally advanced disease is allowed.
3. Patient with bone metastases only
4. Patient has symptomatic CNS metastases; patients with asymptomatic CNS metastases may participate in this trial. The patient must have completed any prior local treatment for CNS metastases ≥ 15 days prior to the start of study treatment (including radiotherapy and/or surgery) and must have completed corticosteroid therapy.
5. Patient has a concurrent malignancy or malignancy within 3 years of study enrollment
6. Patient has received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study
7. Patients who have received chemotherapy or targeted anticancer therapy ≤ 4 weeks (6 weeks for nitrosourea, antibodies or mitomycin-C; 3 weeks for weekly chemotherapy) prior to starting study drug or who have not recovered from side effects of such therapy
8. Patients who have received any continuous or intermittent small molecule therapeutics (excluding monoclonal antibodies) ≤ 5 effective half-lives prior to starting study drug or who have not recovered from side effects of such therapy
9. Patients who have undergone major surgery ≤ 28 days prior to starting study drug or who have not recovered from side effects of such therapy
10. Known diagnosis of human immunodeficiency virus (HIV) infection
11. Patient has a known hypersensitivity to paclitaxel or other products containing Cremophor
12. Patient has a contraindication to use the paclitaxel standard pre-treatment such as corticosteroids
13. Patients with any peripheral neuropathy ≥ CTCAE grade 2
14. Patients with diarrhea ≥ CTCAE grade 2
15. Patient has active cardiac disease
16. Patient has a history of cardiac dysfunction including
17. Patients who are currently receiving treatment with medication with a known risk prolong the QT interval or inducing Torsades de Pointes
18. Patient has poorly controlled diabetes mellitus (HbA1c > 8 %)
19. Other concurrent severe and/or uncontrolled concomitant medical conditions
20. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of LY2780301
21. Patient is currently receiving treatment with drugs known to be substrate of isoenzyme CYP3A4
22. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL)
23. Patient who does not apply effective contraception during the study and through the duration as defined below after the final dose of study treatment.
24. Other experimental treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Phase Ib: recommended phase II dose (RP2D) | Day 28
  To determine the recommended phase II dose (RP2D) of daily LY2780301 when administered orally in combination with weekly intravenous (IV) paclitaxel in HER2-negative, inoperable locally advanced or MBC patients
Phase II: objective response rate (ORR) | until progression assessed up to 18 months
  To estimate the efficacy of daily LY2780301 when administered orally at the RP2D in combination with weekly intravenous (IV) paclitaxel in HER2-negative, inoperable locally advanced or MBC patients, in the overall population and in patients with activation of PI3/AKT/S6 pathway

SECONDARY OUTCOMES:
safety | up to the end of treatment or maximum 6 months
  Type and severity of adverse events according to CTCAE v4.0 up to the end of treatment or maximum 6 months
clinical benefit (CB) | until progression assessed up to 18 months
  The Clinical benefit (CB) is defined as the addition of complete response (CR) + partial response (PR) + Stable disease (SD) > 6 months
progression-free survival (PFS) | until progression assessed up to 18 months
  Date of progression (evaluated according to RECIST V1.1 criteria) or death up to 18 months
pharmacokinetics | D1, D8, D15, D22, D28 post dose
  Pharmacokinetics of LY2780301 and paclitaxel evaluated by plasma concentrations and basic PK parameters

CONTACTS AND LOCATIONS:
Overall Officials: Anthony GONCALVES, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (2):
- France (2):
  - Centre Geroges François Leclerd, Dijon
  - Institut Paoli-Calmettes, Marseille

REFERENCES:
- [Derived] Sabatier R, Vicier C, Garnier S, Guille A, Carbuccia N, Isambert N, Dalenc F, Robert M, Levy C, Pakradouni J, Adelaide J, Chaffanet M, Sfumato P, Mamessier E, Bertucci F, Goncalves A. Circulating tumor DNA predicts efficacy of a dual AKT/p70S6K inhibitor (LY2780301) plus paclitaxel in metastatic breast cancer: plasma analysis of the TAKTIC phase IB/II study. Mol Oncol. 2022 May;16(10):2057-2070. doi: 10.1002/1878-0261.13188. Epub 2022 Mar 30. PMID 35122700
- [Derived] Vicier C, Sfumato P, Isambert N, Dalenc F, Robert M, Levy C, Rezai K, Provansal M, Adelaide J, Garnier S, Guille A, Carbuccia N, Popovici C, Charafe-Jauffret E, Chaffanet M, Birnbaum D, Pakradouni J, Bertucci F, Boher JM, Sabatier R, Goncalves A. TAKTIC: A prospective, multicentre, uncontrolled, phase IB/II study of LY2780301, a p70S6K/AKT inhibitor, in combination with weekly paclitaxel in HER2-negative advanced breast cancer patients. Eur J Cancer. 2021 Dec;159:205-214. doi: 10.1016/j.ejca.2021.09.040. Epub 2021 Nov 12. PMID 34781168
- See also: official web site of the sponsor — http://institutpaolicalmettes.fr